CLINICAL TRIAL: NCT03578627
Title: Psychological/Immunity Studies With Women With Cancer Previously
Brief Title: Stress and Immunity Breast Cancer Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Barbara Andersen, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1992C0350
Record Dates: First submitted 2018-06-19; First posted 2018-07-06 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer Stage II; Breast Cancer Stage III
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assessment-only (No Intervention)
- Intervention (Experimental)
  Interventions: Behavioral: BioBehavioral Intervention

INTERVENTIONS:
Behavioral: BioBehavioral Intervention — Psychological (stress and quality of life), behavioral (health behaviors and compliance), and biologic (neuroendocrine and immune) factors, and pathways by which health outcomes (e.g. disease endpoints-recurrence, disease free interval) might be affected.
  Arms: Intervention

SUMMARY:
An investigative study of the effectiveness of the BioBehavioral Intervention on Stage II/III breast cancer patients. A total of 231 patients were split between an assessment-only control group and an experimental group receiving the Intervention and assessment. The goal of the Intervention is to use psychological, behavioral, and biologic methods with the primary goal of reducing cancer recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Stage II or III breast cancer diagnosis prior to adjuvant therapy

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 1994-05-01 (Actual); Primary Completion 2000-05-31 (Actual); Study Completion 2000-05-31 (Actual)

PRIMARY OUTCOMES:
Recurrence event | Ten years
  Diagnosis of pathologically confirmed breast cancer recurrence
Recurrence time | Ten years
  Time from the day of initial stage II or III breast cancer diagnosis to day of pathology confirmed breast cancer recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Andersen, Principal Investigator — The Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Conley CC, Andersen BL. Lemons to lemonade: Effects of a biobehavioral intervention for cancer patients on later life changes. Health Psychol. 2019 Mar;38(3):206-216. doi: 10.1037/hea0000717. PMID 30762400
- See also: The Jamesline — http://cancer.osu.edu